CLINICAL TRIAL: NCT03266822
Title: T-cell Subsets in Rheumatoid Arthritis Patients on Long-term Anti-TNF or IL6-receptor-blocker Therapy
Status: Completed | Type: Observational
Sponsor: Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: ETT-TUKEB905/PI/09
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control
  Interventions: Other: No intervention
- RA patients on anti-TNF therapy
- RA patients on anti-IL-6R therapy

INTERVENTIONS:
Other: No intervention — Observational study
  Groups: Healthy control

SUMMARY:
Data on the impact of biological therapies, especially of IL6-blocker treatment, on the T-cell phenotype in rheumatoid arthritis (RA) are limited, inconclusive, and mainly involve short-term follow-up.

Here, the investigator prospectively measure the percentages of 15 circulating T-cell subtypes using flow cytometry. The investigators aim to obtained transversal and longitudinal data in 30 anti-TNF responders, 19 secondary anti-TNF-non-responders, 43 IL6R-antagonist-responders before, 8 weeks and, after, at least, 6 months of biological therapy. These are then compared with results obtained in early, untreated RA patients and gender-and-age matched healthy controls.

ELIGIBILITY:
Inclusion Criteria for patients:

* Diagnosis of rheumatoid arthritis classified according to the 2010 ACR/EULAR classification criteria for RA
* Biological treatment with anti-TNF therapy (adalimumab or certolizumab pegol or etanercept or infliximab or golimumab) or anti-IL-6R agent (tocilizumab)

Inclusion Criteria for healthy controls:

* negative history of RA symptoms
* negative status upon detailed physical and laboratory examination including normal CRP and ESR values

Exclusion Criteria:

* other autoimmune comorbidity
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the cross-sectional analysis, 92 RA patients (who had been treated with biological therapy for more than six months) were evaluated.
  As a further control group (healthy controls), we enrolled 30 age- and gender-matched healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Flow cytometry for the assessment of change in T cell subtypes | Before, after 8 weeks and after at least 6 months of the initiation of biological therapy.
  The percentages of 15 circulating T-cell subtypes were measured using flow cytometry.

IPD SHARING:
Plan to Share IPD: Undecided
Upon request

REFERENCES:
- [Derived] Dulic S, Vasarhelyi Z, Sava F, Berta L, Szalay B, Toldi G, Kovacs L, Balog A. T-Cell Subsets in Rheumatoid Arthritis Patients on Long-Term Anti-TNF or IL-6 Receptor Blocker Therapy. Mediators Inflamm. 2017;2017:6894374. doi: 10.1155/2017/6894374. Epub 2017 Oct 25. PMID 29209104